CLINICAL TRIAL: NCT01339975
Title: Level of Expression and Prognostic Value of CXCL4, CXCL4L1 and CXCR3 in Renal Cell Carcinoma
Acronym: ChemoRenCan
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2010/45
Record Dates: First submitted 2011-04-20; First posted 2011-04-21 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Carcinoma; Carcinoma Renal Cell; Kidney Neoplasms; Kidney Diseases; Chemokines
Keywords: Renal Cell Carcinoma; Nephrectomy; Antiangiogenics; Chemokines; Prognostic value; Carcinoma; Carcinoma, Renal Cell; Kidney Neoplasms; Kidney Diseases; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Adenocarcinoma; Urologic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Urologic Diseases; Adjuvants, Immunologic; Physiological Effects of Drugs; Pharmacologic Actions; Biomarkers; Targeted therapies; Surgery
MeSH Terms: conditions — Carcinoma; Carcinoma, Renal Cell; Kidney Neoplasms; Kidney Diseases; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Adenocarcinoma; Urologic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Urologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, urine and tissues
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A. Surgically treated patients: Patients having a radical or partial nephrectomy.
  Interventions: Biological: Biological sample
- Group B. Patients treated with targeted therapies: Patients treated by RCC-directed targeted therapy
  Interventions: Biological: Biological sample

INTERVENTIONS:
Biological: Biological sample — 2 blood samples of 10mL + one urine sample
  * on pre-operative d-1/d, post-operative d1 and d5(+/-2),
  * one month post-operative,
  * at the end of the study in the absence of disease progression or at the date of recurrence or progression if the case arises.
  Groups: Group A. Surgically treated patients
Biological: Biological sample — 2 blood samples of 10mL + one urine sample
  * before starting the therapy
  * at first therapeutic evaluation (2 or 3 months depending on the treatment chosen)
  * at the end of the study or at the date of disease progression.
  Groups: Group B. Patients treated with targeted therapies

SUMMARY:
Despite novel treatment options, Renal Cell Carcinoma (RCC) has been characterized by a constant increase in its mortality and consequently requires an important involvement in translational research.

The aim of this study is to evaluate the interest of CXCL4, CXCL4L1 and CXCR3 as biomarkers in localized, locally advanced or metastatic RCC. Indeed these chemokines have shown anti-angiogenic and anti-tumor properties in experimental models and may be particularly interesting for prognostic and predictive purposes.

DETAILED DESCRIPTION:
Based on a physiopathological rationale, the use of RCC-directed antiangiogenic therapies into clinical practice leads to conclusive results and makes RCC a particularly well-suited tumor type to study factors involved in the angiogenic process. Furthermore the intensive use of targeted therapies in clinical practice raised new questions about their management.

Therefore the identification of new molecular biomarkers is important:

* to improve the precision of prognostic models currently based on clinical, biological or histopathological variables
* to identify high risk patients that could benefit from an adjuvant treatment or a closer postoperative follow-up
* to predict the response to antiangiogenic therapies and therefore identify the drug which is likely to be the most effective within an ever increasing pharmacopeia
* to follow the therapy as precisely as possible, predict or attest the disease progression justifying a therapeutic modification

Low CXCL4, CXCL4L1 and CXCR3 tumor expression levels are associated with bad prognosis factors in RCC. Consequently their interest in RCC is worth being evaluated, in two subgroups : Localized / locally advanced renal cell carcinoma and Metastatic renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with localized, locally advanced or metastatic Renal Cell Carcinoma :

  * having a radical or partial nephrectomy
  * or treated by RCC-directed targeted therapy
* Patients who have signed and dated an informed consent form with the investigator

Exclusion Criteria:

* under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with localized, locally advanced or metastatic Renal Cell Carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2011-06-06 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Prognostic value of the markers of interest (CXCL4, CXCL4L1 et CXCR3) | 3 years
  Prognostic value of the markers of interest (CXCL4, CXCL4L1 et CXCR3) will be evaluated by the association of these markers with time to event occurrence.
  Localized or locally advanced renal cell carcinoma group:
  * local recurrence
  * contralateral recurrence
  * extra-renal distant recurrence (metastatic progression)
  * specific cancer death
  * nonspecific cancer death
  Metastatic renal cell carcinoma group :
  * local recurrence for patients who underwent a nephrectomy
  * contralateral reccurence
  * metastatic progression
  * specific cancer death
  * nonspecific cancer death

SECONDARY OUTCOMES:
Predictive value of therapeutic response | 3 years
  Predictive value of therapeutic response will be assessed for patients receiving systemic therapy. It will be evaluated by the association of markers of interest with the therapeutic response.
  * RECIST criteria: patients showing a complete response or a partial response, will be considered as "responders"
  * The progression of the longest diameter of tumor, the proportion of intra-tumor necrosis (Choi criteria) and +/- the perfusion characteristics of tumor if primitive tumor

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe BERNHARD, Dr, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- University Bordeaux Hospital, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belot A, Grosclaude P, Bossard N, Jougla E, Benhamou E, Delafosse P, Guizard AV, Molinie F, Danzon A, Bara S, Bouvier AM, Tretarre B, Binder-Foucard F, Colonna M, Daubisse L, Hedelin G, Launoy G, Le Stang N, Maynadie M, Monnereau A, Troussard X, Faivre J, Collignon A, Janoray I, Arveux P, Buemi A, Raverdy N, Schvartz C, Bovet M, Cherie-Challine L, Esteve J, Remontet L, Velten M. Cancer incidence and mortality in France over the period 1980-2005. Rev Epidemiol Sante Publique. 2008 Jun;56(3):159-175. doi: 10.1016/j.respe.2008.03.117. Epub 2008 Jun 10. PMID 18547762
- [Background] Raynal G, Bernhard JC. [Premature death from urologic cancer: the kidneys at the forefront]. Prog Urol. 2007 Apr;17(2):260-1. doi: 10.1016/s1166-7087(07)92277-0. No abstract available. French. PMID 17489332
- [Background] Motzer RJ, Mazumdar M, Bacik J, Berg W, Amsterdam A, Ferrara J. Survival and prognostic stratification of 670 patients with advanced renal cell carcinoma. J Clin Oncol. 1999 Aug;17(8):2530-40. doi: 10.1200/JCO.1999.17.8.2530. PMID 10561319
- [Background] Margulis V, Sanchez-Ortiz RF, Tamboli P, Cohen DD, Swanson DA, Wood CG. Renal cell carcinoma clinically involving adjacent organs: experience with aggressive surgical management. Cancer. 2007 May 15;109(10):2025-30. doi: 10.1002/cncr.22629. PMID 17420980
- [Background] Mickisch GH, Garin A, van Poppel H, de Prijck L, Sylvester R; European Organisation for Research and Treatment of Cancer (EORTC) Genitourinary Group. Radical nephrectomy plus interferon-alfa-based immunotherapy compared with interferon alfa alone in metastatic renal-cell carcinoma: a randomised trial. Lancet. 2001 Sep 22;358(9286):966-70. doi: 10.1016/s0140-6736(01)06103-7. PMID 11583750
- [Background] Motzer RJ, Hutson TE, Tomczak P, Michaelson MD, Bukowski RM, Rixe O, Oudard S, Negrier S, Szczylik C, Kim ST, Chen I, Bycott PW, Baum CM, Figlin RA. Sunitinib versus interferon alfa in metastatic renal-cell carcinoma. N Engl J Med. 2007 Jan 11;356(2):115-24. doi: 10.1056/NEJMoa065044. PMID 17215529
- [Background] Escudier B, Eisen T, Stadler WM, Szczylik C, Oudard S, Siebels M, Negrier S, Chevreau C, Solska E, Desai AA, Rolland F, Demkow T, Hutson TE, Gore M, Freeman S, Schwartz B, Shan M, Simantov R, Bukowski RM; TARGET Study Group. Sorafenib in advanced clear-cell renal-cell carcinoma. N Engl J Med. 2007 Jan 11;356(2):125-34. doi: 10.1056/NEJMoa060655. PMID 17215530
- [Background] Escudier B, Pluzanska A, Koralewski P, Ravaud A, Bracarda S, Szczylik C, Chevreau C, Filipek M, Melichar B, Bajetta E, Gorbunova V, Bay JO, Bodrogi I, Jagiello-Gruszfeld A, Moore N; AVOREN Trial investigators. Bevacizumab plus interferon alfa-2a for treatment of metastatic renal cell carcinoma: a randomised, double-blind phase III trial. Lancet. 2007 Dec 22;370(9605):2103-11. doi: 10.1016/S0140-6736(07)61904-7. PMID 18156031
- [Background] Ravaud A, Wallerand H, Culine S, Bernhard JC, Fergelot P, Bensalah K, Patard JJ. Update on the medical treatment of metastatic renal cell carcinoma. Eur Urol. 2008 Aug;54(2):315-25. doi: 10.1016/j.eururo.2008.04.056. Epub 2008 May 5. PMID 18485581
- [Background] Maione TE, Gray GS, Petro J, Hunt AJ, Donner AL, Bauer SI, Carson HF, Sharpe RJ. Inhibition of angiogenesis by recombinant human platelet factor-4 and related peptides. Science. 1990 Jan 5;247(4938):77-9. doi: 10.1126/science.1688470.
- [Background] Jouan V, Canron X, Alemany M, Caen JP, Quentin G, Plouet J, Bikfalvi A. Inhibition of in vitro angiogenesis by platelet factor-4-derived peptides and mechanism of action. Blood. 1999 Aug 1;94(3):984-93. PMID 10419890
- [Background] Lasagni L, Francalanci M, Annunziato F, Lazzeri E, Giannini S, Cosmi L, Sagrinati C, Mazzinghi B, Orlando C, Maggi E, Marra F, Romagnani S, Serio M, Romagnani P. An alternatively spliced variant of CXCR3 mediates the inhibition of endothelial cell growth induced by IP-10, Mig, and I-TAC, and acts as functional receptor for platelet factor 4. J Exp Med. 2003 Jun 2;197(11):1537-49. doi: 10.1084/jem.20021897. PMID 12782716
- [Background] Eisman R, Surrey S, Ramachandran B, Schwartz E, Poncz M. Structural and functional comparison of the genes for human platelet factor 4 and PF4alt. Blood. 1990 Jul 15;76(2):336-44. PMID 1695112
- [Background] Struyf S, Burdick MD, Proost P, Van Damme J, Strieter RM. Platelets release CXCL4L1, a nonallelic variant of the chemokine platelet factor-4/CXCL4 and potent inhibitor of angiogenesis. Circ Res. 2004 Oct 29;95(9):855-7. doi: 10.1161/01.RES.0000146674.38319.07. Epub 2004 Sep 30. PMID 15459074
- [Background] Struyf S, Burdick MD, Peeters E, Van den Broeck K, Dillen C, Proost P, Van Damme J, Strieter RM. Platelet factor-4 variant chemokine CXCL4L1 inhibits melanoma and lung carcinoma growth and metastasis by preventing angiogenesis. Cancer Res. 2007 Jun 15;67(12):5940-8. doi: 10.1158/0008-5472.CAN-06-4682. PMID 17575164
- [Background] Pan J, Burdick MD, Belperio JA, Xue YY, Gerard C, Sharma S, Dubinett SM, Strieter RM. CXCR3/CXCR3 ligand biological axis impairs RENCA tumor growth by a mechanism of immunoangiostasis. J Immunol. 2006 Feb 1;176(3):1456-64. doi: 10.4049/jimmunol.176.3.1456. PMID 16424173
- [Background] Klatte T, Seligson DB, Leppert JT, Riggs SB, Yu H, Zomorodian N, Kabbinavar FF, Strieter RM, Belldegrun AS, Pantuck AJ. The chemokine receptor CXCR3 is an independent prognostic factor in patients with localized clear cell renal cell carcinoma. J Urol. 2008 Jan;179(1):61-6. doi: 10.1016/j.juro.2007.08.148. Epub 2007 Nov 13. PMID 17997430
- [Background] Kattan MW, Reuter V, Motzer RJ, Katz J, Russo P. A postoperative prognostic nomogram for renal cell carcinoma. J Urol. 2001 Jul;166(1):63-7. PMID 11435824
- [Background] Motzer RJ, Bacik J, Murphy BA, Russo P, Mazumdar M. Interferon-alfa as a comparative treatment for clinical trials of new therapies against advanced renal cell carcinoma. J Clin Oncol. 2002 Jan 1;20(1):289-96. doi: 10.1200/JCO.2002.20.1.289. PMID 11773181
- [Background] Zisman A, Pantuck AJ, Wieder J, Chao DH, Dorey F, Said JW, deKernion JB, Figlin RA, Belldegrun AS. Risk group assessment and clinical outcome algorithm to predict the natural history of patients with surgically resected renal cell carcinoma. J Clin Oncol. 2002 Dec 1;20(23):4559-66. doi: 10.1200/JCO.2002.05.111. PMID 12454113
- [Background] Bensalah K, Pantuck AJ, Crepel M, Verhoest G, Mejean A, Valeri A, Ficarra V, Pfister C, Ferriere JM, Soulie M, Cindolo L, De La Taille A, Tostain J, Chautard D, Schips L, Zigeuner R, Abbou CC, Lobel B, Salomon L, Lechevallier E, Descotes JL, Guille F, Colombel M, Belldegrun AS, Patard JJ. Prognostic variables to predict cancer-related death in incidental renal tumours. BJU Int. 2008 Nov;102(10):1376-80. doi: 10.1111/j.1464-410X.2008.07847.x. Epub 2008 Aug 22. PMID 18727618
- [Background] Furniss D, Harnden P, Ali N, Royston P, Eisen T, Oliver RT, Hancock BW; National Cancer Research Institute Renal Clinical Studies Group. Prognostic factors for renal cell carcinoma. Cancer Treat Rev. 2008 Aug;34(5):407-26. doi: 10.1016/j.ctrv.2007.12.008. Epub 2008 Apr 28. PMID 18440705